CLINICAL TRIAL: NCT06414174
Title: Comparison Between Split Septum and Mechanical Valve Needleless Connector in Preventing Central Line-Associated Bloodstream Infections in Very Preterm Babies or Birth Weight <1500 Grams at Cipto Mangunkusumo Hospital Neonatology Unit
Brief Title: Comparison Between Split Septum and Mechanical Valve Needleless Connector in Preterm Babies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Putri Maharani Tristanita Marsubrin, MD, PhD, Neonatologist, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NeedlelessInd
Record Dates: First submitted 2024-05-03; First posted 2024-05-16 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Sepsis, Neonatal
MeSH Terms: conditions — Neonatal Sepsis

STUDY DESIGN:
Intervention Model Description: This study involves two group of participants to receive specific intervention. One of the group will be using split septum mechanism for their needleless connector, while the other group will use mechanical valve mechanism for their needleless connector. Both group will be assessed and monitored closely for the incidence of infection
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Very preterm neonates or birth weight < 1500 gram receiving split septum needleless connector (Active Comparator): Very preterm neonates or birth weight < 1500 gram who needs central line access will use split septum mechanism for their needleless connector
  Interventions: Device: Split septum needleless connector
- Very preterm neonates or birth weight < 1500 gram receiving mechanical valve needleless connector (Active Comparator): Very preterm neonates or birth weight < 1500 gram who needs central line access will use mechanical valve for their needleless connector
  Interventions: Device: Mechanical valve needleless connector

INTERVENTIONS:
Device: Split septum needleless connector — Participants in this study are limited to very preterm neonates or neonates with birth weight under 1500 grams. Split septum mechanism is still widely use in Indonesia, therefore the use of mechanical valve mechanism as needleless connector for central line access in very preterm neonates have never been tested.
  Arms: Very preterm neonates or birth weight < 1500 gram receiving split septum needleless connector
Device: Mechanical valve needleless connector — Participants in this study are limited to very preterm neonates or neonates with birth weight under 1500 grams. Split septum mechanism is still widely use in Indonesia, therefore the use of mechanical valve mechanism as needleless connector for central line access in very preterm neonates have never been tested.
  Arms: Very preterm neonates or birth weight < 1500 gram receiving mechanical valve needleless connector

SUMMARY:
The goal of this clinical trial study is to compare the effectiveness between split septum and mechanical valve needleless connector in very preterm babies (or under 1500 grams)

The main questions it aims to answer are:

* What is the incidence of Central Line-Associated Bloodstream Infections when using a split septum connector?
* What is the incidence of Central Line-Associated Bloodstream Infections when using a mechanical valve connector?
* What is the ratio length of stay between babies with birth weight < 1500 grams who use split septum connector and mechanical valve?
* What is the ratio incidence of mortality due to sepsis of babies with birth weight < 1500 grams who use split septum connector and mechanical valve?

Participants will be observed for two weeks after insertion of central line. They will be taken blood sample for culture and sepsis marker panel.

Researchers will compare split septum group and mechanical valve group to see if there is a central line associated bloodstream infections

ELIGIBILITY:
Inclusion Criteria:

* Preterm neonates with gestational age less than and equal to 32 weeks
* Birth weight less than 1500 gram
* Neonates indicated to use central line access
* Parents are willing to participate in this study and has filled and signed the informed consent letter

Exclusion Criteria:

* Neonates who are previously diagnosed as CLABSI
* Neonates who has other focus of infection that are diagnosed before the recruitment
* Suffer from congenital abnormalities

Ages: 28 Weeks to 32 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2024-08-30 (Actual); Primary Completion 2025-01-14 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
Incidence of Central Line Associated Bloodstream Infection (CLABSI) | From the date of central line insertion until the date of documented infection, whichever came first, assessed up to 30 days
  The incidence of CLABSI are proven by clinical symptoms followed by positive blood culture taken at two different site, consist of peripheral and central site

SECONDARY OUTCOMES:
Length of stay | From the date of admission until the date of discharged or death, which ever comes first, assessed up to 100 days
  The duration which the subject is hospitalized
CLABSI-related mortality | From the date of central line insertion until the date of death, assessed up to 30 days
  Incidence of death because of sepsis in CLABSI participant
All-cause mortality | From the date of admission until the date of death, assessed up to 100 days
  Incidence of death in all participant
Central line days | From the date of central line insertion until the date of death, discharge, or maximum duration of 14 days, whichever comes first
  The duration of central line insertion
Hospitalization cost | From the date of admission until the date of death or discharge, whichever comes first, assessed up to 100 days
  The total cost of hospitalization in each participant

CONTACTS AND LOCATIONS:
Locations (1):
- Cipto Mangunkusumo Hospital, Jakarta Pusat, Jakarta Special Capital Region, Indonesia

IPD SHARING:
Plan to Share IPD: No
The data will not be shared because of the confidentiality agreement stated in the informed consent form

REFERENCES:
- [Background] Muller M, Bryant KA, Espinosa C, Jones JA, Quach C, Rindels JR, Stewart DL, Zangwill KM, Sanchez PJ. SHEA Neonatal Intensive Care Unit (NICU) White Paper Series: Practical approaches for the prevention of central-line-associated bloodstream infections. Infect Control Hosp Epidemiol. 2023 Apr;44(4):550-564. doi: 10.1017/ice.2022.53. Epub 2022 Mar 4. PMID 35241185
- [Background] Jansen SJ, Broer SDL, Hemels MAC, Visser DH, Antonius TAJ, Heijting IE, Bergman KA, Termote JUM, Hutten MC, van der Sluijs JPF, d'Haens EJ, Kornelisse RF, Lopriore E, Bekker V. Central-line-associated bloodstream infection burden among Dutch neonatal intensive care units. J Hosp Infect. 2024 Feb;144:20-27. doi: 10.1016/j.jhin.2023.11.020. Epub 2023 Dec 14. PMID 38103692
- [Background] Urrea Ayala M, Almendral A, Jordan Garcia I, Reyne Vergeli M, Porron R, Llado Maura Y, Limon E, Pujol M; VINCat Pediatric and Neonatal ICU Bacteremia Programme. Central line-associated bloodstream infections (CLABSI) in pediatric and neonatal intensive care units-The VINCat program 2013-2022. Enferm Infecc Microbiol Clin (Engl Ed). 2025 May;43 Suppl 1:S90-S97. doi: 10.1016/j.eimce.2024.09.014. Epub 2025 Mar 12. PMID 40082115
- [Background] Field K, McFarlane C, Cheng AC, Hughes AJ, Jacobs E, Styles K, Low J, Stow P, Campbell P, Athan E. Incidence of catheter-related bloodstream infection among patients with a needleless, mechanical valve-based intravenous connector in an Australian hematology-oncology unit. Infect Control Hosp Epidemiol. 2007 May;28(5):610-3. doi: 10.1086/516660. Epub 2007 Apr 12. PMID 17464926
- [Background] Marschall J, Mermel LA, Fakih M, Hadaway L, Kallen A, O'Grady NP, Pettis AM, Rupp ME, Sandora T, Maragakis LL, Yokoe DS; Society for Healthcare Epidemiology of America. Strategies to prevent central line-associated bloodstream infections in acute care hospitals: 2014 update. Infect Control Hosp Epidemiol. 2014 Jul;35(7):753-71. doi: 10.1086/676533. No abstract available. PMID 24915204
- [Background] Ryder M, deLancey-Pulcini E, Parker AE, James GA. Bacterial transfer and biofilm formation in needleless connectors in a clinically simulated in vitro catheter model. Infect Control Hosp Epidemiol. 2023 Nov;44(11):1760-1768. doi: 10.1017/ice.2023.60. Epub 2023 Apr 24. PMID 37088696
- [Background] Jarvis WR, Murphy C, Hall KK, Fogle PJ, Karchmer TB, Harrington G, Salgado C, Giannetta ET, Cameron C, Sherertz RJ. Health care-associated bloodstream infections associated with negative- or positive-pressure or displacement mechanical valve needleless connectors. Clin Infect Dis. 2009 Dec 15;49(12):1821-7. doi: 10.1086/648418. PMID 19911973
- [Background] Li R, Cao X, Shi T, Xiong L. Application of peripherally inserted central catheters in critically ill newborns experience from a neonatal intensive care unit. Medicine (Baltimore). 2019 Aug;98(32):e15837. doi: 10.1097/MD.0000000000015837. PMID 31393341
- [Background] Westergaard B, Classen V, Walther-Larsen S. Peripherally inserted central catheters in infants and children - indications, techniques, complications and clinical recommendations. Acta Anaesthesiol Scand. 2013 Mar;57(3):278-87. doi: 10.1111/aas.12024. Epub 2012 Dec 17. PMID 23252685
- [Background] Geldenhuys C, Dramowski A, Jenkins A, Bekker A. Central-line-associated bloodstream infections in a resource-limited South African neonatal intensive care unit. S Afr Med J. 2017 Aug 25;107(9):758-762. doi: 10.7196/SAMJ.2017.v107i9.12124. PMID 28875883
- [Background] Nielsen CL, Zachariassen G, Holm KG. Central line-associated bloodstream infection in infants admitted to a level lllneonatal intensive care unit. Dan Med J. 2022 Apr 7;69(5):A05210463. PMID 35485786
- [Background] Zipursky AR, Yoon EW, Emberley J, Bertelle V, Kanungo J, Lee SK, Shah PS; Canadian Neonatal Network Investigators. Central Line-Associated Blood Stream Infections and Non-Central Line-Associated Blood Stream Infections Surveillance in Canadian Tertiary Care Neonatal Intensive Care Units. J Pediatr. 2019 May;208:176-182.e6. doi: 10.1016/j.jpeds.2018.12.011. Epub 2019 Mar 8. PMID 30853200